CLINICAL TRIAL: NCT00661440
Title: Efficacy and Safety of Neramexane Mesylate in Congenital Idiopathic Nystagmus and Acquired Nystagmus: a Randomized, Double-blind, Placebo-controlled, Single Center, Proof of Concept Study Using a Two-period Cross-over Design
Brief Title: Efficacy and Safety Study of Neramexane to Treat Congenital and Acquired Nystagmus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merz Pharmaceuticals GmbH (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: MRZ 92579-0707/1; EudraCT Number 2007-002595-34
Record Dates: First submitted 2008-04-15; First posted 2008-04-18 (Estimated); Last update posted 2009-11-26 (Estimated); Status verified 2009-11

CONDITIONS: Nystagmus, Congenital Idiopathic; Nystagmus, Acquired
MeSH Terms: conditions — Nystagmus, Pathologic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Other)
  Interventions: Drug: Neramexane mesylate
- 2 (Other)
  Interventions: Drug: Neramexane mesylate

INTERVENTIONS:
Drug: Neramexane mesylate — 2 double-blind, cross-over treatment periods of 7 weeks separated by a wash-out phase, up to 75 mg Neramexane mesylate per day
  Other Names: - verum, placebo; - placebo, verum

SUMMARY:
The purpose of this study is to investigate the safety and efficacy of neramexane mesylate in the treatment of congenital idiopathic nystagmus (CIN) in comparison to placebo. In addition, a subgroup of multiple sclerosis (MS) patients suffering from acquired nystagmus will be included; this subgroup will be analyzed in an exploratory manner only.

ELIGIBILITY:
Inclusion Criteria:

* patients with congenital idiopathic nystagmus or acquired nystagmus subsequent to multiple sclerosis
* male or female outpatients
* aged between 18 and 80 years (inclusive) at screening

Exclusion Criteria:

* patients with evidence of neurologic disorders other than CIN such as congenital nystagmus due to albinism or retinal diseases and/or acquired nystagmus (exemption: secondary to MS)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2008-05

PRIMARY OUTCOMES:
Visual acuity | Screening, Baseline, Week 3, 7, 11, 14, 18, and Follow-up

SECONDARY OUTCOMES:
nystagmus intensity, expanded nystagmus acuity function, reading ability, questionnaires, safety parameter

CONTACTS AND LOCATIONS:
Overall Officials: Irene Gottlob, Prof., MD, Principal Investigator — University of Leicester, Leicester, United Kingdom
Locations (1):
- University of Leicester, Leicester Royal Infirmary, Ophthalmology Group, Leicester, United Kingdom